CLINICAL TRIAL: NCT05269498
Title: Navigation Support With Mixed Reality for Surgical Clipping of Cerebral Aneurysms in Adult Patients With CORTEXPLORER MED - a Pilot Stage, Exploratory, First in Human Clinical Investigation
Brief Title: Navigation Support With Mixed Reality With CORTEXPLORER MED
Acronym: CXmed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: cortEXplore GmbH (Industry)
Collaborators: Raffeiner GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CXmed_001
Record Dates: First submitted 2022-02-25; First posted 2022-03-08 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Cranial Aneurysm
Keywords: Neuronavigation; Neurosurgery; Aneurysm; Surgical navigation
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CORTEXPLORER MED (Experimental): Mixed-reality assisted planning of aneurysm clipping with the optical navigation system CORTEXPLORER MED.
  Interventions: Device: CORTEXPLORER MED

INTERVENTIONS:
Device: CORTEXPLORER MED — The CORTEXPLORER MED system is a platform that enables surgical navigation using real-time radiological images of patients. The application software formats patient-specific computed tomography or magnetic resonance images taken before surgery. These are displayed on the screen and through mixed reality from different perspectives (axial, sagittal, coronal, diagonal). Before surgery, the surgeon can then create, save and simulate the course along one or more surgical trajectories. As a visualization aid, the surgeon can also create and edit one or more 3D models of the anatomy. During surgery, the system tracks the position of specific surgical instruments in or on the patient's anatomy and continuously updates the position of the instruments on these images.

SUMMARY:
During the last 15 years, neuronavigation has become an essential neurosurgical tool for pursuing minimal invasiveness and safety. One drawback of such devices is the fact, that the neurosurgeon has to look away from the surgical field onto a dedicated workstation screen. Additionally, the operator is required to transfer this information from the "virtual" environment of the navigation system to the real surgical field - whereas the real patient may be fixated and positioned differently compared to the visualization on the screen.

Mixed-reality may have the potential to support this, by merging data from the real environment with virtual information and vice-versa. In the context of surgical navigation, the main goal of mixed reality systems is to provide a real-time updated 3D virtual model of anatomical details, overlaid on the real surgical field. In this sense, the mixed reality is the process of enrichment of reality with additional virtual contents.

This clinical investigation aims at the collecting of clinical data about the mixed-reality supported planning, the registration accuracy and overall precision of the navigation system and the clinical outcome.

DETAILED DESCRIPTION:
The CORTEXPLORER MED system is a platform that enables surgical navigation using radiological images of patients. The application software reads, formats and merges patient-specific multimodal images such as pre-surgical computed tomography (CT), magnetic resonance imaging (MRI, fMRI) as well as intraoperatively taken fluoroscopic scans. These digital representations of the patient are displayed on a computer screen from different anatomical perspectives (axial, sagittal, coronal, diagonal). Moreover, a 3D digital model can be computed based on the 2D imaging data. Before the operation, the surgeon can create, save, and simulate the course along one or more surgical trajectories. During surgery, the system tracks the position of specific surgical instruments in or on the patient's anatomy and continuously updates their position, which can be displayed on a computer screen or trough mixed reality glasses (Microsoft HoloLens).

Generally, this clinical investigation aims at the collecting of clinical data to indicate the difference between the planning of a neurosurgery without and with the mixed reality feature of CORTEXPLORER MED.

Additionally, clinical data is collected to indicate the difference between the planning of a surgery with the CORTEXPLORER MED and without the system (conventional approach for this indication).

The data from this pilot phase are used for the planning of a larger clinical investigation and for the overall clinical evaluation of the navigation system.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any gender in the age older or eqal 18 years
* Patients who be informed of the nature of the clinical investigation and provide written informed consent
* Patients with a cerebral aneurysm for which surgical clipping is indicated
* Patients with a cerebral aneurysm where clipping is not routinely supported by navigation
* Patients with current (not longer than 4 months) 3D image data of the brain

Exclusion Criteria:

* Patients for whom required imaging is not available
* Patients with ruptured cerebral aneurysm
* Detained patients
* Patients performing mandatory military service / community service
* Patients who refuse to participate in the clinical investigation
* Pregnant or nursing patients
* Patients who are not able to sign the consent form
* Patients who do not speak German
* Patients who are taking part in any other clinical investigations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Estimated trajectory with mixed-reality (without projection of trajectory) | Day 0
  Difference of angle and position of the estimated trajectory with mixed-reality support and without the projected trajectory compared to the pre-operatively defined trajectory.
Estimated trajectory without mixed-reality | Day 0
  Difference of angle and position of the estimated trajectory without mixed reality support (conventional) compared to the pre-operatively defined trajectory.

SECONDARY OUTCOMES:
Estimated trajectory with mixed-reality (with projection of trajectory) | Day 0
  Difference of angle and position of the estimated trajectory with mixed reality support and with the projected trajectory compared to the pre-operatively defined trajectory.
Estimated trajectory with navigation support (planning view) | Day 0
  Difference of angle and position of the estimated trajectory with navigation support (planning view) compared to the pre-operatively defined trajectory.
Estimated trajectory with navigation support (navigation view) | Day 0
  Difference of angle and position of the estimated trajectory with navigation support (navigation view) and with the projected trajectory compared to the pre-operatively defined trajectory.
Planning performance with CORTEXPLORER MED | Day 0, Day 30
  The distance to vessels and the distance from the cranial surface to the target of the post-surgical planning and the initial estimation of the trajectory (conventional approach).
Registration accuracy | Day 0
  The registration accuracy is measured with the navigation software in millimeters
Usability questionnaire | Day 0, Day 30
  Usability questionnaire related to the activities preparation, planning, navigation and post-processing [0 - 5]
Degree of disability or limitation | Day 7
  Degree of disability or limitation in the daily activities of patients after neurological interventions as measured with the Modified Rankin Scale
Intraoperative complications | Day 0
  Severity and occurrence of seizures and bleedings and other intraoperative adverse events
Postoperative complications | Day 1 to Day 7
  Severity and occurrence of seizures and bleedings and other postoperative adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Gmeiner, MD, Principal Investigator — Johannes-Kepler-University, Department of Neurosurgery
Locations (1):
- Kepler Universitätsklinikum, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Homepage of manufacturer — http://www.cortexplore.com